CLINICAL TRIAL: NCT02929719
Title: A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study, Comparing Test Gel, 5% to ACZONE Gel, 5% and Both Active Treatment to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: Study Comparing Test to Aczone 5% and Both to a Placebo Control in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPSG 1518, 1216
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Gel 5% (Experimental): Topical, twice daily on the face for 84 days.
  Interventions: Drug: Test.
- ACZONE Gel 5% (Active Comparator): Topical, twice daily on the face for 84 days
  Interventions: Drug: Aczone Gel 5%
- Placebo Gel (Placebo Comparator): Topical, twice daily on the face for 84 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Test. — gel
  Other Names: dapsone
  Arms: Test Gel 5%
Drug: Aczone Gel 5% — gel
  Other Names: dapsone
  Arms: ACZONE Gel 5%
Drug: Placebo — gel
  Other Names: Vehicle
  Arms: Placebo Gel

SUMMARY:
Therapeutic equivalence and safety study

DETAILED DESCRIPTION:
To evaluate the therapeutic equivalence and safety of Test formulation and marketed Reference Listed Drug (RLD).

To demonstrate the superiority of efficacy of the Test and Reference products over the placebo control in the treatment.

To compare the safety of Test, Reference and Placebo treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 12 and ≤ 40years with a clinical diagnosis of acne vulgaris
* Subjects must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment (IGA) (per Table 1 below)

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1134 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion count | baseline to week 12 (study day 84)
Change in non-inflammatory lesion count | baseline to week 12 (study day 84)

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No